CLINICAL TRIAL: NCT03319797
Title: Prospective, Multicenter, Single-arm Phase III Clinical Trial to Evaluate the Efficacy and Safety of NOVOCART® Inject Plus in the Treatment of Cartilage Defects of the Knee
Brief Title: NOVOCART® Inject Plus for Cartilage Defects of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tetec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-1624
Record Dates: First submitted 2017-06-14; First posted 2017-10-24 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Cartilage Defects of the Knee
Keywords: Autologous chondrocyte transplantation ACT

STUDY DESIGN:
Intervention Model Description: Prospective, Multicenter, Single-arm Phase III
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with NOVOCART® Inject plus (Other): Treatment with NOVOCART® Inject plus (Autologous chondrocyte transplantation)
  Interventions: Drug: NOVOCART® Inject plus

INTERVENTIONS:
Drug: NOVOCART® Inject plus — Treatment with NOVOCART® Inject plus (Autologous chondrocyte implantation)

SUMMARY:
Prospective, Multicenter, Single-arm Phase III Clinical Trial to Evaluate the Efficacy and Safety of NOVOCART® Inject plus in the Treatment of Cartilage Defects of the Knee. The primary objective of this trial is to demonstrate efficacy of NOVOCART® Inject plus for the treatment of cartilage defects of the knee based on the Knee injury and Osteoarthritis Outcome Score (KOOS) responder rate 24 month after transplantation.

DETAILED DESCRIPTION:
The present study is a prospective, multicenter, single-arm phase III clinical trial to evaluate the efficacy and safety of NOVOCART® Inject plus in the treatment of patients with focal cartilage defects of the knee (medial or lateral femoral condyle or tibial plateau, trochlea or patella). The study will include adult patients between 18 and 65 years of age and pediatric patients (14 to 17 years) with closed epiphysis.

A total of 96 patients will be enrolled in the NOVOCART® Inject plus trial at about 20 clinical study sites in Europe. It is expected that each study site will enroll 3 to 9 patients.

The trial will consist of three phases (including screening, treatment and follow-up phase) with a maximum duration of 5 years and 4 months.

The treatment with NOVOCART® Inject plus requires 2 surgeries. During the first surgery autologous chondrocytes for transplant production will be harvested arthroscopically, then NOVOCART® Inject plus will be transplanted during a second surgery about 3 to 4 weeks later. In general, NOVOCART® Inject plus transplantation can be performed arthroscopically. However, depending on the defect localization, mini-arthrotomy may be indicated.

Eligibility will be assessed preoperatively at visit 1 (screening) and (up to a maximum of 3 months later) intraoperatively during the first arthroscopy (visit 2). During visit 2, cartilage biopsy samples will be taken from eligible patients and sent to TETEC AG for NOVOCART® Inject plus manufacturing. Transplantation will then be performed during a second arthroscopy 3 to 4 weeks later (visit 3).

All patients will be followed up for 5 years post NOVOCART® Inject plus transplantation with assessments at 3, 6, 12, 18, 24, 36, 48 and 60 months as outlined in the schedule of events and treatment at the end of this synopsis.

NOVOCART® Inject plus will be applied in conjunction with a rehabilitation program according to the rehabilitation regimen defined in the clinical study protocol.

The primary and secondary endpoints will be assessed after a follow-up of 24 month post NOVOCART® Inject plus transplantation (primary analysis). Long-term data will be assessed after an additional 3 years follow-up (follow-up analysis).

An interim analysis of efficacy and safety data will be performed when 63 patients (66% of the planned number of patients) are evaluable for the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 and ≤ 65 years old at screening. Pediatric patients (14 to 17 years) with closed epiphysis may be included in selected countries. Closure of the distal femoral epiphysis of the target knee needs to be confirmed by MRI or x-ray.
2. Patients with focal articular cartilage defect(s) of the femoral condyle (medial or lateral), the trochlea, the patella or the tibial plateau (medial or lateral) of the knee.
3. Patient has one or two defects in the target knee with a defect-grade of III or IV according to the International Cartilage Repair Society (ICRS) classification or grade III or IV ICRS classification of osteochondritis dissecans lesions (ICRS-OCD).
4. If the patient has only one grade III or IV defect, the size of the defect is ≥ 4 and ≤ 12 cm2 post debridement. If the patient has two grade III or IV cartilage defects the total defect size is ≥ 4 and ≤ 12 cm2 post debridement. The defects must be located on different, knee joint areas and both cartilage defects are to be treated with NOVOCART® Inject plus.
5. Patient has an intact, well contained chondral structure surrounding the defect (i.e. no diffusely thinned-out cartilage surface) and an articulating joint surface opposite to the defect(s) to be treated (≤ Grade I ICRS or ICRS-OCD classification).
6. Patient has intact menisci in the target knee; a maximum of 50% resection per meniscus is allowed. Completely healed meniscal transplants are accepted.
7. Patient has a stable knee joint or sufficiently reconstructed ligaments and no patella malalignment or a sufficiently corrected patella malalignment. Ligament repair is accepted, if performed before, during or within 6 weeks after NOVOCART® Inject plus transplantation. Correction of patella malalignment must be performed before or during NOVOCART® Inject plus transplantation.
8. Patient has free range of motion (ROM) of the affected knee joint or ≤ 10° of active extension and flexion loss (compared to the other knee).
9. Patient has a baseline score of < 65/100 in the overall KOOS (KOOS5).
10. Only for female patients of childbearing potential (sexually mature, pre-menopausal and not surgically sterile): the patient is willing to use a medically accepted method of contraception until the day of NOVOCART® Inject plus transplantation.
11. Patient is willing and able to give written informed consent to participate in the study and to comply with all follow-up visits and assessments and the postoperative rehabilitation program.

Intraoperative inclusion criteria:

At visit 2, the following inclusion criteria from visit 1 need to be confirmed; all criteria must be answered with "yes" before the patient is considered eligible for the study:

1. Patient is not pregnant as confirmed by urine pregnancy test before arthroscopy
2. Patients with focal articular cartilage defect(s) of the femoral condyle (medial or lateral), the trochlea, the patella or the tibial plateau (medial or lateral) of the knee.
3. Patient has one or two defects in the target knee with a defect-grade of III or IV according to the International Cartilage Repair Society (ICRS) classification or grade III or IV ICRS classification of osteochondritis dissecans lesions (ICRS-OCD).
4. If the patient has only one grade III or IV defect, the size of the defect is ≥ 4 and ≤ 12 cm2 post debridement. If the patient has two grade III or IV cartilage defects the total defect size is ≥ 4 and ≤ 12 cm2 post debridement. The defects must be located on different knee joint areas and both cartilage defects are to be treated with NOVOCART® Inject plus.
5. Patient has an intact intact, well-contained chondral structure surrounding the defect (i.e. no diffusely thinned out cartilage surface) and an articulating joint surface opposite to the defect(s) to be treated (≤ Grade I ICRS or ICRS-OCD classification).
6. Patient has intact menisci in the target knee; a maximum of 50% resection per meniscus is allowed. Completely healed meniscal transplants are accepted.

Exclusion Criteria:

1. Patient is unable to undergo magnetic resonance imaging (MRI).
2. Patient has grade II cartilage defects according to the ICRS or ICRS-OCD classification in the target knee.
3. Patient has more than 2 grade III or IV cartilage defects according to the ICRS or ICRS-OCD classification in the target knee.
4. The cartilage defects (ICRS or ICRS-OCD grade I or III or IV) affect more than 3 out of 6 joint areas1 of the target knee.
5. Patient had a prior biologic reconstructive procedure (e.g. microfracture, mosaicplasty, chondrocyte transplantation) in the target knee at a location different from the defect location to be treated in the study. Prior biologic reconstructive procedures are accepted, if the previously treated defect is the same defect that is planned to be treated with NOVOCART® Inject plus (i.e. the prior method has failed) and these procedures were performed ≥ 24 months prior to screening visit 1.
6. Patient had other prior surgical interventions interfering with the assessment of the NOVOCART® Inject plus treatment. Prior diagnostic arthroscopies with debridement and lavage are acceptable.
7. Patients with subchondral bone defects more than 2 mm deep (after resection of affected bone) unless adjuvant defect filling will be performed before or during NOVOCART® Inject plus transplantation.
8. Patient has degenerative joint disease in the target knee as determined by Kellgren and Lawrence grade >2.
9. Patient has chronic inflammatory arthritis and/or infectious arthritis.
10. Patient has joint space narrowing > 1/3 in the target knee when compared to the other knee or < 3 mm joint space.
11. Patient has malalignment (valgus- or varus-deformity) in the target knee. Note: In suspected cases, the mechanical axis must be established radiographically by complete leg imaging in standing position and in anteriorposterior (a.p.) or rather posterioranterior (p.a.) projection. The Mikulicz line is not allowed to deviate more than 5 mm of the eminentia intercondylaris. If alignment is necessary, surgery has to be performed before, during or within 6 weeks after NOVOCART® Inject plus transplantation.
12. Patient has arthrofibrosis in the target knee.
13. Patient has diffuse chondromalacia (grade 1 'softening or swelling of cartilage' according to Outerbridge allowed).
14. Patient has metabolic arthropathies (e.g. gout, pseudo-gout)
15. Patient has bilateral lower limb pain or low back pain.
16. Patient has a known systemic connective tissue disease.
17. Patient has a current uncontrolled diabetes.
18. Patient has a known history of autoimmune disease.
19. Patient has a known history of immunological suppressive disorder or is taking immunosuppressants.
20. Patient is currently systemically or intra-articularly taking steroids and/or has used steroids within the last 30 days prior to screening visit 1.
21. The patient has a history of Human Immunodeficiency Virus (HIV)/ Acquired Immune Deficiency Syndrome (AIDS), Human T cell lymphotropic virus (HTLV), syphilis (Treponema pallidum) or active hepatitis B or C (HCV) infection with verified antigens. Patients with a cured hepatitis B or C infection and/or verified antibodies are not excluded.
22. The patient has a history of borreliosis.
23. The patient has an active systemic or local (at the site of surgery) infection, eczematization or inflammable skin alterations.
24. Patient has a known history of cancer within the past 5 years.
25. Patient has a known history of osteoporosis, uncontrolled primary hyperparathyroidism or hyperthyroidism, chronic renal failure or prior pathological fractures independent of the genesis.
26. Patient has any degenerative muscular or neurological condition that would interfere with evaluation of outcome measures including but not limited to Parkinson's disease, amyotrophic lateral sclerosis (ALS), or multiple sclerosis (MS).
27. Patient has a body mass index (BMI) > 35 kg/m2.
28. Patient is a woman who is pregnant or lactating.
29. Patient is currently participating, or has participated in any other clinical study within 3 months prior to screening visit 1.
30. Patient has known current or recent history of illicit drug or alcohol abuse or dependence.
31. Patient has psychiatric or cognitive impairment that, in the opinion of the investigator, would interfere with the patient's ability to comply with the study requirements, e.g., Alzheimer's disease.
32. Patient has a known intolerance to any constituents of NOVOCART® Inject plus.
33. Patient has comorbidities preventing the patient from undergoing surgery
34. Patient has any other condition, which, in the opinion of the investigator, would make the patient unsuitable for the study.

Intraoperative exclusion criteria:

At visit 2, the following exclusion criteria from visit 1 need to be confirmed; all criteria must be answered with "no" before the patient is considered eligible for the study:

1. Patient has grade II cartilage defects according to the ICRS or ICRS-OCD classification in the target knee.
2. Patient has more than 2 grade III or IV cartilage defects according to the ICRS or ICRS-OCD classification in the target knee.
3. The cartilage defects (ICRS or ICRS-OCD grade I or III or IV) affect more than 3 out of 6 joint areas2 of the target knee.
4. Patients with subchondral bone defects more than 2 mm deep (after resection of affected bone) unless adjuvant defect filling will be performed before or during NOVOCART® Inject plus transplantation.
5. Patient has arthrofibrosis in the target knee.
6. Patient has diffuse chondromalacia (grade 1 'softening or swelling of cartilage' according to Outerbridge allowed).

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Responder rate based on the Knee injury and Osteoarthritis Outcome Score (KOOS5). The KOOS score ranges from 0 to 100 (100 indicating no symptoms and 0 indicating extreme symptoms). | 24 month
  Responder rate based on the Knee injury and Osteoarthritis Outcome Score (KOOS5) defined as the average of the 5 subscale scores (ensuring identical weight from all subscales) at the 24 months follow-up assessment. The KOOS5 responder rate is defined as the proportion of patients with ≥ 10 points improvement in the KOOS5 from baseline to the 24 months visit.

SECONDARY OUTCOMES:
Change in the KOOS5 | 24 month
  Change in the KOOS5 from baseline
Change in the 5 individual subscores of the KOOS | 24 month
  Change in the 5 individual subscores of the KOOS from baseline
Change in the International Knee Documentation Committee (IKDC) subjective score. The IKDC score ranges from 0 to 100, with 100 indicating the absence of symptoms and higher levels of functioning. | 24 month
  Change in the International Knee Documentation Committee (IKDC) subjective score from baseline
Change in EQ-5D-5L. The components are the EQ-5D-5L index ranging from <0 (worse than dead) to 1 (full health) and a visual analogue scale with the end points of 0 (worst health) and 100 (best health). | 24 month
  Change from baseline in the EQ-5D-5L questionnaire
Change in activity level/ functional status. Patient questionnaire on activity (sporting habits) and functional status (degree of restriction in general), no score provided. | 24 months
  Change from baseline in activity level/ functional status
Patient satisfaction with treatment. Patients will be asked 4 questions (with 3 answer options each) related to their treatment satisfaction, no score provided. | 24 month
  Patient satisfaction with treatment after NOVOCART® Inject plus transplantation (questionnaire)
Change in the grading according to the IKDC surgeons part | 24 month
  Change from baseline in the grading according to the IKDC surgeons part
Morphological assessment of the Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score | 24 month
  In vivo performance measured by the morphological assessment of the Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score in a subgroup of 48 patients
Biochemical MR assessment by T2 mapping | 24 month
  Biochemical MR assessment by T2 mapping in a subgroup of 48 patients
Time to treatment failure | 24 month
  Treatment failure is defined as all surgical re-interventions affecting the closed surface of the transplant and/or require additional cartilage repair modalities on the target defect.
Treatment failure rate | 24 month
  Treatment failure is defined as all graft-related conditions requiring surgical re-intervention
Treatment-related adverse events (AEs) | 24 month
  Treatment-related adverse events (AEs) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Niemeyer, MD, Principal Investigator — Orthopaedic Surgery Munich
Locations (20):
- Czechia (6):
  - Orthopedic department of Hospital of Rudolf and Stefanie Benešov, Benešov
  - Clinic of traumatology Úrazová nemocnice Brno, Brno
  - NH Hospital, a.s., Department of Orthopaedics, Hořovice Hospital, Hořovice
  - Orthopaedic Department of Faculty Hospital Ostrava, Ostrava
  - Orthopaedic department of Hospital pardubice, Hospital of Pardubice Region, Pardubice
  - Clinic of child and adult orthopaedics and traumatology 2nd Medical faculty Charles University and FH Motol, Prague
- Germany (3):
  - University Hospital Freiburg, Department for Orthopaedics and Trauma Surgery, Freiburg im Breisgau
  - Orthodoc MVZ orthopaedics and surgery at medical center Sophienhof GmbH, Kiel
  - Orthopaedic Surgery Munich, Munich
- Hungary (6):
  - Uzsoki Hospital, Budapest
  - Szabolcs-Szatmár-Bereg County Hospitals and University Teaching Hospital, Jósa András Teaching Hospital, Nyíregyháza
  - Bács-Kiskun County Hospital, Teaching Hospital of Faculty of Medicine of University of Szeged, Szeged
  - Szegedi Tudományegyetem Ortopédiai Klinika, Szeged
  - Jász-Nagykun-Szolnok County Hetényi Géza Hospital - Clinic, Traumatology, Szolnok
  - Kastélypark Clinic, Tata
- Lithuania (3):
  - "Ortopedijos technika", PLC, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda university hospital, Klaipėda
- Switzerland (2):
  - Orthopedics "at Rhy", Basel
  - Centrum for orthopedics & sports, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Niemeyer P, Hanus M, Belickas J, Laszlo T, Gudas R, Fiodorovas M, Cebatorius A, Pastucha M, Hoza P, Magos K, Izadpanah K, Pasa L, Vasarhelyi G, Sisak K, Mohyla M, Farkas C, Kessler O, Kybal S, Spiro R, Kohler A, Kirner A, Trattnig S, Gaissmaier C. Treatment of Large Cartilage Defects in the Knee by Hydrogel-Based Autologous Chondrocyte Implantation: Two-Year Results of a Prospective, Multicenter, Single-Arm Phase III Trial. Cartilage. 2022 Jan-Mar;13(1):19476035221085146. doi: 10.1177/19476035221085146. PMID 35354310